CLINICAL TRIAL: NCT02120118
Title: A Phase II Clinical Trial Evaluating the Safety and Efficacy of Combination of Hyperthermia and Concurrent Chemoradiotherapy (CCRT) in Treatment Failure Solid Tumors
Brief Title: Combination of Hyperthermia and Concurrent Chemoradiotherapy (CCRT) in Treatment Failure Solid Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Taiwan FDA asked for seperating this protocol into one disease site per protocol.
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140101D; 20140101D (Other: ShinKongHospital)
Record Dates: First submitted 2014-03-17; First posted 2014-04-22 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2014-10

CONDITIONS: Solid Tumors
Keywords: Treatment failure
MeSH Terms: interventions — Radiation; Diathermy; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation; Hyperthermia; Chemotherapy (Experimental): Patients will be treated with radiotherapy with 50Gy/22fx/6 weeks, plus hyperthermia 42℃ ± 0.5℃ for 40 minutes within 2hr after irradiation, once a week since the 1st week of radiation for a total of 6 times. The regimen of concurrent chemotherapy will cisplatin 30mg/m2 and taxotere 20mg/m2 per week for 6 weekly cycles.
  Interventions: Radiation: Radiation; Other: Hyperthermia; Drug: Cisplatin; Drug: Taxotere

INTERVENTIONS:
Radiation: Radiation — 2Gy/5fx/week for a subtotal of 40Gy/20fx/4 weeks, followed by reduced-field boost with 10Gy/2fx/2 weeks (5Gy once a week during 5th and 6th week), totalling 50Gy/22fx/6 weeks.
Other: Hyperthermia — 42℃ ± 0.5℃ for 40 minutes within 2hr after irradiation, once a week since the 1st week of radiation for a total of 6 times
Drug: Cisplatin — 30mg/m2
Drug: Taxotere — 20mg/m2

SUMMARY:
The primary goals of hyperthermia combined with chemotherapy/radiotherapy on treatment failure solid tumors are tumor response rate, while secondary goals are rates of acute and late adverse effects, local control rate, distant metastasis rate, progression-free rate and overall survival rate.

DETAILED DESCRIPTION:
The goal of this study is to conduct a phase II clinical trial evaluating the safety and efficacy of combination of low temperature (40-43℃ range) hyperthermia and concurrent chemoradiotherapy (CCRT) in treatment failure solid tumors. There are 3 reasons of conducting this clinical trial. Firstly, it has been demonstrated that hyperthermia can enhance the efficacy of chemotherapy, radiotherapy or chemoradiotherapy in various cancers, with acceptable safety profiles. Secondly, the salvage outcomes for treatment failure solid tumors were frustrated. Thermal enhancement ratio (TER) was observed when using hyperthermia combining radiotherapy or chemotherapy. This strategy should be investigated in its efficacy in treating those failing from previous standard treatment and maybe several times of salvage therapy. Thirdly, biologically reciprocal complementation between hyperthermia, chemotherapy and radiotherapy was observed. The reason may be complicated, including theories involving hypoxia, immunomodulation and reperfusion … etc. If the immunity microenvironment could be improved by addition of hyperthermia, an unexpected survival benefit as compared with the literature may be potentially demonstrated from this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 20-85 years, with ECOG performance 0-2.
2. Treatment failure solid tumor(s), with histologically or clinically confirmed recurrence or progression after primary treatment of either single modality of surgery, chemotherapy or radiotherapy or any combinations.
3. Complete surgical excision is NOT feasible as salvage treatment for the recurrent or progressive tumor(s), or the patient does NOT agree to receive the surgical procedure.
4. Salvage radiotherapy is possible, and a total dose of 50Gy/22fx is considered tolerable.
5. Measurable lesions by image examinations or endoscopy within 2 months.
6. The distribution of the lesions of interest does NOT exceed 20cm range.
7. The patient can tolerate implementation of cisplatin and taxotere weekly therapy, with respect to hematopoietic status, renal function, liver function, allergy and other potential adverse effects.

Exclusion Criteria:

1. Re-irradiation of 50Gy/22fx is considered NOT tolerable.
2. Future tumor response to treatment in this study is NOT possibly evaluated using image examinations or endoscopy.
3. The patient is participating in other clinical trials.
4. Future regular clinical follow-up is NOT possible.
5. The patient has large-area metallic implants within hyperthermia field (not including metallic hemoclips with small area and few numbers).
6. The patient has pacemakers.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Tumor response rate | 12 weeks
  To estimate the tumor response rate (complete response + partial response; CR + PR; according to RECIST criteria version 1.1).

SECONDARY OUTCOMES:
Adverse events | up to 12 weeks
  To estimate rates of each grade adverse events (CTCAE, version 4.0) which is possibly, probably, or definitely related to treatment and which occurs within 3 months from the start of radiation combined with hyperthermia and chemotherapy.
Late adverse events | up to 1 years
  To estimate rates of late adverse events.
Time to Disease Progression | up to 5 years
  To estimate the local control rate, distant metastasis rate and progression-free rate for patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan